CLINICAL TRIAL: NCT00229268
Title: FOXA2 Expression in Adipose Tissue of Human Subjects With Obesity/Insulin-Resistance
Brief Title: Research on the Nature, Diagnosis, and Treatment of Obesity and Diabetes
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: MST-0513
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Insulin Resistance; Obesity
Keywords: Healthy Volunteers
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether the level of FOXA2 expression in fat tissue is a biomarker of insulin resistance. To test this hypothesis, we will perform euglycemic-hyperinsulinemic clamps in normal and obese human subjects to calculate insulin sensitivity, and see if insulin sensitivity correlates with the FOXA2 expression in subcutaneous fat.

DETAILED DESCRIPTION:
The investigators at Rockefeller University Hospital are engaged in research on the nature, diagnosis and treatment of obesity and diabetes. The investigators are trying to find out why insulin, a blood sugar lowering hormone that is released by the pancreas following a meal, does not work effectively in individuals with obesity or type 2 diabetes. The investigators have recently discovered a protein in fat cells of obese mice that helps fat cells to take up and break down sugar from the blood. This protein (called FOXA2) also prevents the generation of more fat cells. FOXA2 is only present in obese mice, but absent from fat stores of lean animals. Insulin can stimulate the production of FOXA2 in fat cells. Furthermore, the levels of FOXA2 protein correlate with the degree of blood insulin levels. In this study, we are would like to determine whether FOXA2 is also produced in fat cells of humans, and if its level correlates with the degree of obesity and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals
2. Age 21-45 years old
3. BMI: either < 25, or 30-35, or > 40
4. All patients must be willing and able to sign an informed consent form -

Exclusion Criteria:

1. Chronic illnesses other the than mild forms of illnesses related to obesity, such as hypertension, hyperlipidemia, and others, that do not require medical treatment
2. Diabetes mellitus previously diagnosed as per subject report or an abnormal 2 hour OGTT at screening
3. Chronic drug treatment for any medical condition
4. Active weight reduction of more than 7 pounds in the last 3 months
5. History of bleeding or blood clotting disorders
6. Subjects with hemoglobin <8.5 gm/dl
7. Changes in smoking habits for the last 6 months
8. Current pregnancy or current breast-feeding in women
9. Allergic reaction to local anesthetics
10. History of anaphylaxis or anaphylactic-like reactions
11. Tendency to form scars (keloids) easily
12. Irregular menses
13. HIV and hepatitis B or C positive subjects -

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers of different BMI classifications
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2005-09; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Stoffel, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States